CLINICAL TRIAL: NCT04367675
Title: Phase 1b Study of INO-5401 Alone or INO-5401 in Combination With INO-9012 Followed by Electroporation in Adult Cancer and Non-Cancer Patients With BRCA1 or BRCA2 Mutations
Brief Title: INO 5401 Vaccination in BRCA1/2 Mutation Carriers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 842686, UPCC 06019
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: BRCA1/2 Mutation
MeSH Terms: interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- INO-5401 (Experimental): Participants receive INO-5401 vaccine, followed by electroporation, on Day 1, Week 4, Week 8, and Week 12
  Interventions: Drug: INO-5401; Device: Cellectra 2000
- INO-5401 and INO-9012 (Experimental): Participants receive INO-5401 and INO-09012 vaccine, followed by electroporation, on Day 1, Week 4, Week 8, and Week 12
  Interventions: Drug: INO-5401; Drug: INO-9012; Device: Cellectra 2000

INTERVENTIONS:
Drug: INO-5401 — INO-5401 contains genes which are active in human cancers (hTERT, PMSA, and WNT1) and are felt to be good targets for the immune system both people who have had cancer or for those at increased risk of getting cancer.
Drug: INO-9012 — INO-9012 contains the gene for IL12, a part of your body's immune system. It is possible that adding this to INO-5401 will increase the immune response to the vaccine.
  Arms: INO-5401 and INO-9012
Device: Cellectra 2000 — The device will deliver a small electric charge through 5 needles to increase the amount of the study vaccine taken up by the muscle.

SUMMARY:
The research study is being conducted to test an experimental vaccine to potentially prevent cancer for people with BRCA1 or BRCA2 mutations. This study will test if the vaccine is safe (without significant side effects) and test a new way of administering vaccines. It will also test whether the vaccine activates your immune system.

ELIGIBILITY:
Cohort A Inclusion Criteria:

1. Signed and dated IRB approved informed consent.
2. Females and males age 18+.
3. Documented carrier of a pathogenic or likely pathogenic mutation in BRCA1 or BRCA2.
4. Diagnosis of invasive breast cancer, invasive ovarian cancer, pancreatic cancer (apart from neuroendocrine) or prostate cancer with completion of adjuvant therapy and no clinical evidence of disease according to standard of care.
5. Minimum of 2 clear sites on the skin to allow for injection.
6. ECOG performance status of 0.
7. Normal ECG or ECG without clinically significant findings and which does not require clinical action.
8. Normal bone marrow, hepatic, and renal function.
9. Females who are post-menopausal only.
10. Male subjects with reproductive potential must be willing to use a condom with female partners of reproductive potential and their female sexual partners should use an additional highly effective method of birth control. This is required from screening through 24 weeks after the last dose of immunotherapy.
11. Able and willing to comply with all study procedures.

Cohort B Inclusion Criteria

1. Signed and dated IRB approved informed consent.
2. Females and males age 18+.
3. Documented carrier of a pathogenic or likely pathogenic mutation in BRCA1 or BRCA2.
4. With or without prior prophylactic (but not therapeutic) mastectomy or salpingo-oophorectomy.
5. Minimum of 2 clear sites on the skin to allow for injection.
6. ECOG performance status of 0.
7. Normal ECG or ECG without clinically significant findings and which does not require clinical action.
8. Normal bone marrow, hepatic, and renal function.
9. Females who are post-menopausal only.
10. Male subjects with reproductive potential must be willing to use a condom with female partners of reproductive potential and their female sexual partners should use an additional highly effective method of birth control. This is required from screening through 24 weeks after the last dose of immunotherapy.
11. Able and willing to comply with all study procedures.

Cohort A Exclusion Criteria

1. Previous treatment with INO-5401 or IL-12 containing therapy, or any other DNA immunotherapy.
2. Prior history of invasive cancer other than those listed above. History of localized superficial non-melanoma skin cancers, melanoma in situ, cervical intraepithelial neoplasia, or breast ductal carcinoma in situ is allowed.
3. Pregnant or breast-feeding subjects.
4. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation; continued participation in an observational study is allowed.
5. Cardiac pre-excitation syndromes.
6. Prior major surgery within 4 weeks of first study treatment.
7. Presence of acute or chronic bleeding or clotting disorder that would contraindicate intramuscular injections or use of blood thinners within 2 weeks of first study treatment.
8. Any concurrent condition requiring the continued or anticipated use of systemic steroids or immunosuppressive therapy. All systemic corticosteroids must be discontinued at least 4 weeks prior to first study treatment.
9. History of clinically significant disease or other immunosuppressive disease.
10. HIV infection.
11. Known history of hepatitis B and/or hepatitis C with active viral replication.
12. Receipt of any blood product within 2 weeks before signing ICF.
13. Administration of any vaccine, except influenza vaccine, within 4 weeks of the first study treatment. Administration of influenza vaccine within 2 weeks of first study treatment.
14. Presence of metal implants or implantable medical device within 5 cm of the planned site of injection/EP including a cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the intended deltoid injection site, unless deemed acceptable by a cardiologist.
15. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
16. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.
17. Any other conditions judged by the investigator that would limit the evaluation of the subject.

Cohort B Exclusion Criteria

1. Previous treatment with INO-5401 or IL-12 containing therapy, or any other DNA immunotherapy.
2. Prior history of invasive cancer other than those listed above. History of localized superficial non-melanoma skin cancers, melanoma in situ, cervical intraepithelial neoplasia, or breast ductal carcinoma in situ is allowed.
3. Pregnant or breast-feeding subjects.
4. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation; continued participation in an observational study is allowed.
5. Cardiac pre-excitation syndromes.
6. Prior major surgery within 4 weeks of first study treatment.
7. Presence of acute or chronic bleeding or clotting disorder that would contraindicate intramuscular injections or use of blood thinners within 2 weeks of first study treatment.
8. Any concurrent condition requiring the continued or anticipated use of systemic steroids or immunosuppressive therapy. All systemic corticosteroids must be discontinued at least 4 weeks prior to first study treatment.
9. History of clinically significant disease or other immunosuppressive disease.
10. HIV infection.
11. Known history of hepatitis B and/or hepatitis C with active viral replication.
12. Receipt of any blood product within 2 weeks before signing ICF.
13. Administration of any vaccine, except influenza vaccine, within 4 weeks of the first study treatment. Administration of influenza vaccine within 2 weeks of first study treatment.
14. Presence of metal implants or implantable medical device within 5 cm of the planned site of injection/EP including a cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the intended deltoid injection site, unless deemed acceptable by a cardiologist.
15. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
16. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.
17. Any other conditions judged by the investigator that would limit the evaluation of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | for 2 years after last dose of study treatment
  Dose-limiting toxicities will be classified by system organ class (SOC), preferred term (PT), severity, and relationship to Study Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinayak S, Cecil DL, Disis ML. Vaccines for breast cancer prevention: Are we there yet? Mol Aspects Med. 2024 Aug;98:101292. doi: 10.1016/j.mam.2024.101292. Epub 2024 Jul 10. No abstract available. PMID 38991631